CLINICAL TRIAL: NCT01949246
Title: Analysis of Circulating Biomarkers in Predicting Response to Cardiac Resynchronization Therapy (CRT) With Biventricular Pacing in Patients With Congestive Heart Failure (BIOCRT)
Brief Title: Biomarkers to Predict CRT Response in Patients With HF (BIOCRT)
Acronym: BIOCRT
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jagmeet Singh, Jagmeet P Singh, M.D. Ph.D., Massachusetts General Hospital
Other Study IDs: 2007P001921
Record Dates: First submitted 2013-09-04; First posted 2013-09-24 (Estimated); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Heart Failure
Keywords: Biomarkers
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CRT patients: Patients undergoing CRT device implantation
- Healthy patients: Healthy controls

SUMMARY:
The prospective study aims:

1. To determine the role and mechanism of biomarkers for prediction of response to CRT
2. To determine the role of biomarkers and their effect on left ventricular remodeling in patients undergoing CRT.

DETAILED DESCRIPTION:
Cardiac resynchronization therapy (CRT) with biventricular pacing has emerged as a novel treatment for congestive heart failure (CHF) not responsive to optimal drug therapy. CRT is associated with significant improvements in hemodynamics and functional status of patients with CHF. The physiologic effect of CRT is achieved via placing electrical leads in the right and left ventricular walls, and synchronizing ventricular contraction. Over time, this leads to ventricular wall reverse remodeling, and sustained improvements in left ventricular ejection fraction (EF).

Currently, the indications for CRT include end-stage heart failure class II-IV with an EF < 35%, and a QRS duration > 120ms. The QRS duration is used as an indicator of the degree of ventricular electromechanical dyssynchrony, however, a growing number of studies have postulated its inability to predict response to therapy. As a result, other measures of mechanical dyssynchrony are being sought to guide therapy. The vast majority of these studies have examined clinical, cardiac, electrocardiographic, and device-specific indices, however, a widely accepted predictor of response to CRT is lacking.

CRT results in electromechanical synchrony, leading to an improved ejection fraction, exercise tolerance, and reduction of symptoms. Although electrical re-synchronization and intra-procedural hemodynamic improvement are achieved after the device is implanted, the sustained clinical improvement is likely due to ventricular reverse remodeling. A major issue with CRT is that approximately a third of patients receiving devices do not achieve improved clinical or functional status, and fail to undergo changes in ventricular geometry, and ventricular remodeling. It remains unknown whether this is due to abnormalities in the factors involved in lead placement or procedural strategies, geometric remodeling, alterations in cardiac energy metabolism, supply of energy (i.e. coronary blood flow), or inappropriate/inadequate microvascular proliferation.

This study will evaluate a series of biochemical markers implicated in pathophysiology of heart failure, in predicting response to CRT with biventricular pacing.

ELIGIBILITY:
Inclusion Criteria:

* Study participant with an approved indication for a CRT or CRT-D system.

  1. New York Heart Association (NYHA) Class II, III, or IV Heart Failure unresponsive to drug therapy.
  2. EF < 35%.
  3. QRS width > 120 ms.
* Study participant receiving optimal medical therapy including ACE inhibitor or Angiotensin Receptor Blocker (ARB), Beta-Blocker, and Diuretic.
* Study participants with a history of significant congestive decompensation events within the last 12 months.

Exclusion Criteria:

* NYHA Class I Heart Failure.
* Co morbidities (e.g., cancer), which may limit lifespan < 6 months.
* Severe aortic stenosis (valve area < 1.0 cm2).
* Study participants that received cardiac surgery or intervention (i.e. coronary artery bypass grafting (CABG), valve surgery, angioplasty, arthrectomy) within the preceding 90 days.
* Study participants with moderate to severe chronic obstructive pulmonary disease (COPD), defined as needing chronic oxygen therapy or recent hospitalization (within 30 days) for COPD flare up.
* Concurrent pregnancy.
* Study participants with primary pulmonary hypertension.
* Study participants on continuous or intermittent infusion therapy for heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Outpatient or inpatient heart failure patients scheduled for CRT implantation
Sampling Method: Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2007-09 (Actual); Primary Completion 2016-01-01 (Actual); Study Completion 2016-01-01 (Actual)

PRIMARY OUTCOMES:
MACE | 2 years
  death, HF hospitalization, left ventricular assist device, heart transplant

SECONDARY OUTCOMES:
CRT clinical response | 6 months
  For the definition of a positive response to CRT, patients will be classified according to the HF Clinical Composite Score (CCS). Responders will be defined as those with improved CCS from baseline to 6 month follow-up. Those not meeting this criterion will be considered nonresponders. An outcome panel consisting of two cardiologists will determine the clinical response of each subject based on review of the medical record. If there is disagreement in the assessment of either baseline or follow-up CCS amongst the two cardiologists, a third cardiologist will adjudicate the case.

CONTACTS AND LOCATIONS:
Overall Officials: Jagmeet P Singh, Principal Investigator — Massachussetts General Hospital; Quynh A Truong, MD MPH, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Truong QA, Januzzi JL, Szymonifka J, Thai WE, Wai B, Lavender Z, Sharma U, Sandoval RM, Grunau ZS, Basnet S, Babatunde A, Ajijola OA, Min JK, Singh JP. Coronary sinus biomarker sampling compared to peripheral venous blood for predicting outcomes in patients with severe heart failure undergoing cardiac resynchronization therapy: the BIOCRT study. Heart Rhythm. 2014 Dec;11(12):2167-75. doi: 10.1016/j.hrthm.2014.07.007. Epub 2014 Jul 8. PMID 25014756
- [Derived] Ajijola OA, Chatterjee NA, Gonzales MJ, Gornbein J, Liu K, Li D, Paterson DJ, Shivkumar K, Singh JP, Herring N. Coronary Sinus Neuropeptide Y Levels and Adverse Outcomes in Patients With Stable Chronic Heart Failure. JAMA Cardiol. 2020 Mar 1;5(3):318-325. doi: 10.1001/jamacardio.2019.4717. PMID 31876927
- [Derived] Bakos Z, Chatterjee NC, Reitan C, Singh JP, Borgquist R. Prediction of clinical outcome in patients treated with cardiac resynchronization therapy - the role of NT-ProBNP and a combined response score. BMC Cardiovasc Disord. 2018 Apr 24;18(1):70. doi: 10.1186/s12872-018-0802-8. PMID 29699498